CLINICAL TRIAL: NCT04214054
Title: Maxillary Sinus Lift With and Without Self Hardening Biphasic Calcium Phosphate and Simultaneous Implant Placement
Brief Title: Maxillary Sinus Lift With and Without Self-hardening Biphasic Calcium Phosphate.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCP for maxillary sinus lift
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Maxillary Sinus Augmentation
Keywords: maxillary sinus lift; Piezosurgery; Grafting materials

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled clinical trial and the participants were allocated randomly into two equal groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moldable self-hardening biphasic calcium phosphate graft (Experimental): Easy graft, a moldable osteocondutive allograft formed of 60% hydroxylapatite and 40% β-tricalcium phosphate (Easy-graft, Sunstar, Gruidor, Degradable solutions AG, Swizerlard).
  Interventions: Other: Moldable self-hardening biphasic calcium phosphate graft
- No graft material (Placebo Comparator)
  Interventions: Procedure: No graft material placed - Blood Clot only

INTERVENTIONS:
Other: Moldable self-hardening biphasic calcium phosphate graft — Incision was performed in the canine area then a full thickness mucoperiosteal flap was elevated and exposure of the lateral aspect of the maxillary sinus. Osteotomy of the buccal window was performed using the piezosurgery device followed by meticulous dissection of the sinus membrane. Drilling the site were implants were to be placed, guided by the preformed surgical stent. Implants of appropriate size were torqued to engage the apical aspect of the implant recipient site. The sinus was augmented with moldable self-hardening biphasic calcium phosphate. Repositioning and suturing of the flap using 3-0 black silk suture material.
  Arms: Moldable self-hardening biphasic calcium phosphate graft
Procedure: No graft material placed - Blood Clot only — A pyramidal full thickness mucoperiosteal flap was performed distal to the canine area with a crestal incision located palatally in the edentulous area and vertical extension of the incision to the buccal vestibule using Bard Parker blade number 15. The flap was reflected exposing the alveolar bone. Lateral window was performed and the sinus membrane was elevated using piezo surgery. Drilling at the sites where implants were to be placed was done using Neobiotech implant drilling Kit. Implants. Implants were placed in a self-tapping fashion using a torque wrench. Flaps were replaced back and sutured using 3-0 black silk suture material.
  Arms: No graft material

SUMMARY:
This study was carried out to compare the outcome of sinus lift without grafting material, versus the use of moldable, self hardening calcium phosphate biomaterials with simultaneous implant placement.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled clinical trial, the study population consisted of 20 patients with missing maxillary posterior teeth and residual bone height 5-7mm. The sample was selected conveniently according to a list of inclusion and exclusion criteria, the participants were allocated randomly into two equal groups. All patients had sinus lift using piezosurgery device with simultaneous implant placement. In group I, blood clot was the only filling material. In group II, moldable, self-hardening calcium phosphate was the filling material. Clinical and radiographic evaluations were done through 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients having missing posterior maxillary teeth
* The vertical height between the floor of the maxillary sinus and the alveolar crest ranged between 5 and 7mm,
* Free from maxillary sinus pathologies
* Adequate oral hygiene
* Acceptable interarch space for the prosthesis

Exclusion Criteria:

* Patients with systemic diseases that directly affect the surgical procedure and/ or the healing of the bone
* immunocompromised status
* Alcoholism
* psychiatric disorders
* Parafunctional habits

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-13 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | 1 week
  Pain was assessed through on a 10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Wound healing | 1 week
  The presence of alveolar osteitis (dry socket) will be determined clinically using BLUM'S criteria. Wound healing was assessed and recorded depending on the absence or presence of dehiscence, every opening along the incision will be recorded as dehiscence , dental tweezers will be used to identify it.
Radiographic Evaluation | 6 months
  Cone beam computed tomography (CBCT) was done. The apparatus and the settings were kept the same during all the preoperative scans to evaluate the amount of vertical bone height gained, the change of bone density and the marginal bone loss postoperatively.
Implant stability | 6 months
  Examining implant stability was done using Osstell (Osstell co. Swedan). It is a noninvasive and easy-to-use system to determine implant stability and to assess the process of osseointegration.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa A. El Sadek, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Ahmed A. A. Sharara, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Magda M Saleh, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Nevien Shawky, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Mazor Z, Horowitz RA, Del Corso M, Prasad HS, Rohrer MD, Dohan Ehrenfest DM. Sinus floor augmentation with simultaneous implant placement using Choukroun's platelet-rich fibrin as the sole grafting material: a radiologic and histologic study at 6 months. J Periodontol. 2009 Dec;80(12):2056-64. doi: 10.1902/jop.2009.090252. PMID 19961389
- [Background] Del Fabbro M, Testori T, Francetti L, Weinstein R. Systematic review of survival rates for implants placed in the grafted maxillary sinus. Int J Periodontics Restorative Dent. 2004 Dec;24(6):565-77. PMID 15626319
- [Background] Cha HS, Kim A, Nowzari H, Chang HS, Ahn KM. Simultaneous sinus lift and implant installation: prospective study of consecutive two hundred seventeen sinus lift and four hundred sixty-two implants. Clin Implant Dent Relat Res. 2014 Jun;16(3):337-47. doi: 10.1111/cid.12012. Epub 2012 Nov 15. PMID 23157674